CLINICAL TRIAL: NCT07275047
Title: Comparison of Ultrasound Guided Serratus Posterior Superior Intercostal Plane Block Versus Paravertebral Block for Postoperative Analgesia After Thoracotomy
Brief Title: Analgesic Efficacy of SPSIP Block Versus Paravertebral Block Following Thoracotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, Assoc Prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 13
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Post-thoracotomy Pain
Keywords: Post-thoracotomy pain; Serratus posterior superior intercostal plane block; Paravertebral Block; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIP (Active Comparator): Participants in this arm will receive an ultrasound-guided Serratus Posterior Superior Intercostal Plane Block. The block will be performed preoperatively with the patient in the appropriate position. A local anesthetic solution will be injected between the serratus posterior superior muscle and the intercostal muscles under real-time ultrasound guidance. The technique aims to achieve postoperative analgesia by providing sensory blockade across targeted thoracic dermatomes. No additional regional block will be performed in this group.
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block
- Group Paravertebral (Active Comparator): Participants in this arm will receive an ultrasound-guided thoracic paravertebral block. The block will be performed preoperatively with the patient in the appropriate position. Under real-time ultrasound guidance, a local anesthetic solution will be injected into the thoracic paravertebral space at the planned level to achieve unilateral somatic and sympathetic nerve blockade. This intervention is intended to provide postoperative analgesia following thoracotomy. No additional regional block will be administered in this group.
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: Serratus Posterior Superior Intercostal Plane Block — Ultrasound-guided regional anesthesia technique performed between the serratus posterior superior muscle and intercostal muscles.
  Other Names: SPSIP Block
  Arms: Group SPSIP
Procedure: Thoracic Paravertebral Block — Ultrasound-guided injection of local anesthetic into the thoracic paravertebral space to provide unilateral analgesia.
  Other Names: Paravertebral Block
  Arms: Group Paravertebral

SUMMARY:
Thoracotomy causes severe postoperative pain that may impair respiratory function and increase complications. This study compares the postoperative analgesic effectiveness of the serratus posterior superior intercostal plane (SPSIP) block and the paravertebral block in patients undergoing thoracotomy. The aim is to determine whether the newly described serratus posterior superior intercostal plane block can serve as a safe and effective alternative to established techniques.

DETAILED DESCRIPTION:
Thoracotomy often causes strong postoperative pain because the ribs, muscles, nerves, and pleura are affected during surgery. This pain can make it difficult for patients to breathe well and may increase the chance of lung problems. Paravertebral block is a well-known method for reducing pain after thoracic surgery, but it can sometimes lead to side effects such as low blood pressure or complications related to deeper needle placement.

The serratus posterior superior intercostal plane block is a newer ultrasound-guided technique. In this method, local anesthetic is injected between the serratus posterior superior muscle and the intercostal muscles. Early studies suggest that it may provide wide pain relief, but its effectiveness specifically in thoracotomy patients has not yet been studied.

This randomized study aims to compare the pain-relieving effects of the serratus posterior superior intercostal plane block with those of the paravertebral block after thoracotomy. The goal is to find out whether this new block can be a safe and effective option for postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo thoracotomy
* ASA physical status I-III according to the American Society of Anesthesiologists classification
* Able to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Declines or is unable to provide informed consent
* Allergy or hypersensitivity to local anesthetics or opioids
* Known or suspected coagulopathy
* Infection at the injection site
* History of thoracic surgery
* Severe cardiovascular disease
* Hepatic or renal failure
* Pregnant, suspected pregnancy, or breastfeeding

Significant neurological or psychiatric disorder that may interfere with study participatio

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative 24-Hour PCA Opioid Consumption | Postoperative 24 hours
  Total amount of opioid delivered by the patient-controlled analgesia (PCA) device during the first 24 hours after surgery, recorded in milligrams (mg).

SECONDARY OUTCOMES:
NRS Pain Scores at Rest and Movement | 2, 4, 8, 16, 24, and 48 hours postoperatively
  Numeric Rating Scale (NRS) (0-10) pain scores at rest and during movement or coughing at predefined postoperative hours.
QoR-15 Recovery Score | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.]
  The investigators will use the Turkish version of Quality of Recovery (QoR) / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  Able to breathe easily Been able to enjoy food Feeling rested Have had a good sleep Able to look after personal toilet and hygiene unaided Able to communicate with Getting support from hospital doctors and nurses Able to return to work or usual home activities Feeling comfortable and in control Having a feeling of general well-being
  PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) Moderate pain Severe pain Nausea or vomiting Feeling worried or anxious Feeling sad or depressed
Chronic Pain Assessment | 3 months postoperatively
  Pain status using the Brief Pain Inventory (BPI) via telephone follow-up.
  General Scoring: The BPI comprises the Pain Severity and Pain Interference subscales. Each item is scored on a 0 (None/No interference) to 10 (Worst imaginable/Completely disabling) numerical scale. Higher scores indicate a worse clinical outcome. Subscale scores are calculated by taking the arithmetic mean of relevant items.
  1. Pain Severity Subscale (4 Items): Assesses pain intensity over the last 24 hours. (0-10) What is your pain level right now What was your pain at its least in the last 24 hours What was your pain at its worst in the last 24 hours What was your pain on average in the last 24 hours
  2. Pain Interference Subscale (7 Items): Assesses the degree to which pain interferes with daily functioning Questions: The patient rates how much pain interfered with: (0-10) General activity Mood Walking ability Normal work Relations with people Sleep Enjoyment of life
Rescue Analgesic Requirement | Postoperative 0-48 hours
  Number of patients requiring rescue analgesia (IV meperidine 0.5 mg/kg) and total dose administered when NRS ≥ 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayman EO, Brennan TJ. Incidence and severity of chronic pain at 3 and 6 months after thoracotomy: meta-analysis. J Pain. 2014 Sep;15(9):887-97. doi: 10.1016/j.jpain.2014.06.005. Epub 2014 Jun 23. PMID 24968967
- [Background] Wildgaard K, Ravn J, Kehlet H. Chronic post-thoracotomy pain: a critical review of pathogenic mechanisms and strategies for prevention. Eur J Cardiothorac Surg. 2009 Jul;36(1):170-80. doi: 10.1016/j.ejcts.2009.02.005. PMID 19307137
- [Background] Mehta S, Jen TTH, Hamilton DL. Regional analgesia for acute pain relief after open thoracotomy and video-assisted thoracoscopic surgery. BJA Educ. 2023 Aug;23(8):295-303. doi: 10.1016/j.bjae.2023.05.001. Epub 2023 Jun 22. No abstract available. PMID 37465231
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Akin AN, Yildiz Y, Alver S, Ciftci B. Continuous serratus posterior superior intercostal plane block for postoperative analgesia management in the patient who underwent right atrial mass excision: a case report. BMC Anesthesiol. 2024 Apr 25;24(1):159. doi: 10.1186/s12871-024-02535-4. PMID 38664657
- [Background] Yildirim Y, Parlar Kilic S, Eyigor S, Eyigor C, Yildirim Y, Karaman E, Oyur Celik G, Uyar M. Validity and reliability of Turkish version of the Brief Pain Inventory-Short Form for patients with chronic nonmalignant pain. Agri. 2019 Nov;31(4):195-201. doi: 10.14744/agri.2019.25901. PMID 31741339